CLINICAL TRIAL: NCT00289770
Title: A Double Blind Randomised, Comparative Study of the Immunogenicity and Reactogenicity of Three Different Lots of GlaxoSmithKline Biologicals' Combined Hepatitis A - Hepatitis B Vaccine When Administered in Healthy Adults
Brief Title: Long-term Immune Persistence of GSK Biologicals' Combined Hepatitis A & B Vaccine Injected According to a 0,1,6 Mth Schedule in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100551 (EXT Y11); 100552 (EXT Y12) (Other: GSK); 100553 (EXT Y13) (Other: GSK); 100554 (EXT Y14) (Other: GSK); 100555 (EXT Y15) (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: TWINRIX™ ADULT; Hepatitis A; Hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — twinrix

ARMS (3):
- Group A (Experimental): Was vaccinated with Lot A in the primary study.
  Interventions: Biological: Twinrix™
- Group B (Experimental): Was vaccinated with Lot B in the primary study.
  Interventions: Biological: Twinrix™
- Group C (Experimental): Was vaccinated with Lot C in the primary study.
  Interventions: Biological: Twinrix™

INTERVENTIONS:
Biological: Twinrix™ — Intramuscular injection, 3 doses

SUMMARY:
The aim of this study is to evaluate the long-term persistence of hepatitis A and B antibodies at Years 11, 12, 13, 14 and 15 after subjects received their first dose of a 3 dose primary vaccination schedule of combined hepatitis A/hepatitis B vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

This protocol posting deals with objectives & outcome measures of the extension phase at Year 11-15.

DETAILED DESCRIPTION:
This is a long-term follow-up study at Years 11, 12, 13, 14 and 15 after primary vaccination with GSK Biologicals' hepatitis A/hepatitis B vaccine (three-dose schedule with 3 different lots). To evaluate the long-term antibody persistence, volunteers will be bled at Years 11, 12, 13, 14 and 15 after the first vaccine dose of the primary vaccination course to determine their anti-HAV and anti-HBs antibody concentrations.

No additional subjects will be recruited in the course of this extension study. If a subject has become seronegative for anti-HAV antibodies or lost anti-HBs seroprotection concentrations at the long-term blood sampling time point (i.e. Years 11, 12, 13, 14 or 15), he/ she will be offered an additional vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had consented to participate in the long-term follow-up studies at the previous long-term blood sampling time points
* Written informed consent will have been obtained from each subject. before the blood sampling visit of each year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-11-01; Primary Completion 2004-12-20 (Actual); Study Completion 2004-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Damme P, Leroux-Roels G, Crasta P, Messier M, Jacquet JM, Van Herck K. Antibody persistence and immune memory in adults, 15 years after a three-dose schedule of a combined hepatitis A and B vaccine. J Med Virol. 2012 Jan;84(1):11-7. doi: 10.1002/jmv.22264. Epub 2011 Nov 3. PMID 22052690
- [Background] Van Damme P, Leroux-Roels G, Law B, Diaz-Mitoma F, Desombere I, Collard F, Tornieporth N, Van Herck K. Long-term persistence of antibodies induced by vaccination and safety follow-up, with the first combined vaccine against hepatitis A and B in children and adults. J Med Virol. 2001 Sep;65(1):6-13. PMID 11505437
- [Background] Van Herck K, Leroux-Roels G, Van Damme P, Srinivasa K, Hoet B. Ten-year antibody persistence induced by hepatitis A and B vaccine (Twinrix) in adults. Travel Med Infect Dis. 2007 May;5(3):171-5. doi: 10.1016/j.tmaid.2006.07.003. Epub 2006 Sep 20. PMID 17448944
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 100551 (EXT Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100551 (EXT Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100551 are summarised with studies 100552, 100553, 100554, and 100555 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 100551 (EXT Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100551 (EXT Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100551 (EXT Y11) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who came back at a follow-up, did not necessarily come back at an earlier timepoint. Therefore amount of subjects who completed the previous timepoint does not always correspond with amount of subjects who entered follow-up. As Year 15 has enrolled the most subjects, baseline measures are given for Year 15, to be as complete as possible.
Groups:
- Twinrix Group: Subjects who were vaccinated with either Lot 1, Lot 2 or Lot 3 of Twinrix in the primary study according to a 0, 1, 6-Month schedule
Period: Year 11
Arm/Group | Twinrix Group
Started | 37
Completed | 37
Not Completed | 0
Period: Year 12
Arm/Group | Twinrix Group
Started | 40
Completed | 40
Not Completed | 0
Period: Year 13
Arm/Group | Twinrix Group
Started | 37
Completed | 37
Not Completed | 0
Period: Year 14
Arm/Group | Twinrix Group
Started | 43
Completed | 43
Not Completed | 0
Period: Year 15
Arm/Group | Twinrix Group
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Twinrix Group
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.4 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis A (Anti-HAV) Antibody Concentrations Equal to or Above Cut-off Value
Description: Cut-off value was defined as 15 milli-international units per milliliter (mIU/mL). This was considered as seropositivity.
Time Frame: Years 11, 12, 13, 14 and 15
Population: Analysis was performed on the long-term (LT) According-To-Protocol (ATP) cohort for immunogenicity, which included subjects who returned at a particular blood sampling timepoint, were in the ATP immunogenicity cohort in the primary study and for whom serology results were available for that particular timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 31
Participants
  Year 11: number analyzed (Participants) | 25
  Year 11 | 25
  Year 12: number analyzed (Participants) | 28
  Year 12 | 28
  Year 13: number analyzed (Participants) | 23
  Year 13 | 23
  Year 14: number analyzed (Participants) | 24
  Year 14 | 24
  Year 15 | 31

2. Primary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above Cut-off Values
Description: Cut-off values were defined 3.3 mIU/mL for the in-house anti-HBs assay and 6.2 mIU/mL for the ChemiLuminescence ImmunoAssay, which was also considered as seropositivity, and 10 mIU/mL.
Time Frame: Years 11, 12, 13, 14 and 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 31
Participants
  Year 11 3.3 mIU/mL: number analyzed (Participants) | 25
  Year 11 3.3 mIU/mL | 23
  Year 12 3.3 mIU/mL: number analyzed (Participants) | 28
  Year 12 3.3 mIU/mL | 25
  Year 13 3.3 mIU/mL: number analyzed (Participants) | 23
  Year 13 3.3 mIU/mL | 20
  Year 14 3.3 mIU/mL: number analyzed (Participants) | 24
  Year 14 3.3 mIU/mL | 21
  Year 14 6.2 mIU/mL: number analyzed (Participants) | 24
  Year 14 6.2 mIU/mL | 21
  Year 15 6.2 mIU/mL | 28
  Year 11 10 mIU/mL: number analyzed (Participants) | 25
  Year 11 10 mIU/mL | 23
  Year 12 10 mIU/mL: number analyzed (Participants) | 28
  Year 12 10 mIU/mL | 25
  Year 13 10 mIU/mL: number analyzed (Participants) | 23
  Year 13 10 mIU/mL | 20
  Year 14 10 mIU/mL: number analyzed (Participants) | 24
  Year 14 10 mIU/mL | 21
  Year 15 10 mIU/mL | 28

3. Primary Outcome: Anti-HAV and Anti-HBs Antibody Concentrations
Description: Concentrations are expressed as geometric mean concentrations (GMCs) in mIU/mL.
  The laboratory assay was changed from Year 13 to Year 14 to in-house ELISA and at Year 15 to CLIA for anti-HBs GMCs.Thus for the sake of bridging, blood samples corresponding to Year 14 previously tested with ELISA were re-tested with CLIA (Year 14*).
Time Frame: Years 11, 12, 13, 14 and 15
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 31
mIU/mL
  Year 11 anti-HAV: number analyzed (Participants) | 25
  Year 11 anti-HAV | 680.3 [453.8 to 1019.9]
  Year 12 anti-HAV: number analyzed (Participants) | 28
  Year 12 anti-HAV | 602.7 [420.8 to 863.2]
  Year 13 anti-HAV: number analyzed (Participants) | 23
  Year 13 anti-HAV | 601.5 [408.7 to 885.4]
  Year 14 anti-HAV: number analyzed (Participants) | 24
  Year 14 anti-HAV | 524.7 [368.7 to 746.5]
  Year 15 anti-HAV | 610.7 [443.1 to 841.6]
  Year 11 anti-HBs: number analyzed (Participants) | 25
  Year 11 anti-HBs | 458.9 [257.4 to 817.8]
  Year 12 anti-HBs: number analyzed (Participants) | 28
  Year 12 anti-HBs | 475.8 [284.4 to 795.9]
  Year 13 anti-HBs: number analyzed (Participants) | 23
  Year 13 anti-HBs | 163.3 [99.7 to 267.3]
  Year 14 anti-HBs: number analyzed (Participants) | 24
  Year 14 anti-HBs | 149.1 [94.8 to 234.5]
  Year 14* anti-HBs: number analyzed (Participants) | 24
  Year 14* anti-HBs | 242.8 [127.0 to 464.3]
  Year 15 anti-HBs | 210.9 [121.5 to 366.2]

4. Primary Outcome: Anti-HBs Antibody Concentrations
Description: Subjects who lost seroprotective concentrations for anti-HBs (< 10 mIU/mL) at any of the LT follow-up timepoints received an additional dose of Engerix after year 15.
  Two subjects were eligible for this after Year 11.
  3.29 in the table means a concentration of < 3.3 mIU/mL.
  As the concentration was calculated per subject no mean concentration was calculated and also no measure of dispersion.
Time Frame: at Year 11, pre-additional vaccine, after additional dose of Engerix
Population: Analysis was performed on the long-term (LT) Total Vaccinated Cohort in subjects who were eligible for an additional dose. This included all subjects who had received at least one dose of the study vaccine in the primary study and who returned for the blood sampling timepoint and who had serology results for anti-HAV and anti-HBs available.
Measure: Number; unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
mIU/mL
  subject 1 Year 11 | 3.29
  subject 2 Year 11 | 3.29
  subject 1 before additional dose | 3.29
  subject 2 before additional dose | 14.5
  subject 1 after additional dose | 6548.1
  subject 2 after additional dose | 554.0

5. Primary Outcome: Number of Subjects, Receiving an Additional Vaccination of Engerix, With an Anamnestic Response
Description: Anamnestic response was assessed in subjects receiving an additional vaccine dose of Engerix. Two subjects were found eligible at Year 11 for this additional vaccine dose.
  Anamnestic response was defined as:
  * post-additional vaccination anti-HBs concentration >= 10 mIU/mL in subject seronegative before additional dose.
  * 4-fold increase post-additional dose compared to pre-additional vaccine time point.
Time Frame: 30 days post additional dose of Engerix
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
Participants | 2

6. Primary Outcome: Number of Subjects With Solicited Local and General Symptoms Assessed
Description: Solicited local symptoms were pain, redness and swelling. Solicited general symptoms were fatigue, fever, gastrointestinal, headache.
Time Frame: During the 4-day follow-up period after additional vaccination with Engerix
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
Participants
  Pain | 0
  Redness | 0
  Swelling | 0
  Fatigue | 1
  Fever | 0
  Gastrointestinal | 1
  Headache | 0

7. Primary Outcome: Number of Subjects With Unsolicited Symptoms
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30-day follow-up period after additional Engerix vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
Participants | 1

8. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject
Time Frame: During the 30-day follow-up period after additional Engerix vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
Participants | 0

9. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Determined by the Investigator to Have a Causal Relationship to Primary Vaccination or Due to Lack of Vaccine Efficacy
Description: as for outcome 8
Time Frame: up to Year 11, 12, 13, 14, 15
Population: Analysis was performed on the long-term (LT) Total Vaccinated Cohort, this included all subjects who had received at least one dose of the study vaccine in the primary study and who returned for the blood sampling time-point and who had serology results for anti-HAV and anti-HBs available.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group
Number analyzed (Participants) | 50
Participants
  Year 11: number analyzed (Participants) | 37
  Year 11 | 0
  Year 12: number analyzed (Participants) | 40
  Year 12 | 0
  Year 13: number analyzed (Participants) | 37
  Year 13 | 0
  Year 14: number analyzed (Participants) | 43
  Year 14 | 0
  Year 15 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected up to Year 15. Other adverse events were collected within 4-days after additional vaccination (solicited) and 30-days after additional vaccination (unsolicited).
Description: As the number of subjects differs for SAEs at the different timepoints the maximum number has been taken for the amount of subjects at risk.
Arm/Group | Twinrix Group
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=2)
Fatigue (General disorders) | 1
Gastrointestinal (General disorders) | 1
Heaviness sensation above eyes (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following complete retesting and reanalysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.